CLINICAL TRIAL: NCT06760208
Title: Korean Post-marketing Surveillance for Prevenar 20
Brief Title: A Study to Learn More About Prevenar 20 Once it is Out in the Korean Market
Status: Not yet recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7471038
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Pneumococcal Immunization; Safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pneumococcal 20-valent conjugate vaccine: Subjects aged 6 weeks or older who have been administered Pneumococcal 20-valent conjugate vaccine as per approved product label.
  Interventions: Biological: Pneumococcal 20-valent conjugate vaccine

INTERVENTIONS:
Biological: Pneumococcal 20-valent conjugate vaccine — For intramuscular use only. One dose (0.5 mL) of Pneumococcal 20-valent conjugate vaccine should be administered intramuscularly, preferably in the deltoid muscle, with care to avoid injection into or near nerves and blood vessels.

SUMMARY:
The purpose of this study is to understand the safety of Prevenar 20 (Pneumococcal 20-valent conjugate vaccine) once it is out in the Korean market. Prevenar 20 will be given to participants aged 6 weeks or older in Republic of Korea.

This study is seeking for participants who are:

* Infant, children and adolescents aged 6 weeks to under 18 years or adult who are 18 years or older
* Prescribed Prevenar 20 by their physician as per approved product label

All participants in this study will receive Prevenar 20 vaccine.

1 dose (0.5 mL) of Prevenar 20 will be given into a muscle, preferably to the shoulder muscle.

We will look at the experiences of people receiving the study medicine. This will help us see if the study medicine is safe.

Participants will take part in this study for 28 days. During this time, study doctor collects the data of subjects to understand the safety of study medicine. There is no strict fixed visit schedule. If subjects are unable to visit the study clinic 28 days after Prevenar 20 vaccine was given then the safety information will be collected by telephone or e-mail.

DETAILED DESCRIPTION:
The study design will reflect the actual management of subjects in routine clinical practice. The study will be performed by continuous registration method. Investigators enroll subjects who receive Prevenar 20 (Pneumococcal 20-valent conjugate vaccine) for the first time after the start of the study.

Data can be collected at routine scheduled and/or unscheduled visits. There is no mandatory fixed visit schedule. Investigator collects the data of subjects from the time of the subject's first dose of study drug to a minimum of 28 days following administration of study drug, to evaluate the safety of study drug and records the information in each subject's Case Report Form.

As no additional visits or tests are required for this study, the data specified in this protocol may not be collected from all subjects.

Endpoint

* Frequency and proportion of solicited systemic reactions occurring from Day 1 through Day 7 after vaccination, where Day 1 is the day of vaccination.
* Frequency and proportion of solicited local reactions occurring from Day 1 through Day 10 days after vaccination, where Day 1 is the day of vaccination.
* Frequency and proportion of Adverse Events (AEs), Adverse Drug Reactions (ADRs), Serious Adverse Events (SAEs), Serious Adverse Drug Reactions (SADRs), Unexpected AEs, Unexpected ADRs, Unexpected SAEs, and Unexpected SADRs throughout the surveillance period
* Frequency and proportion of Adverse Events Special Interest (AESI) throughout the surveillance period

  * Invasive Pneumococcal Disease

All assessments are performed as part of normal clinical practice or standard practice guidelines for the subject population and healthcare provider specialty in the countries where this non-interventional study is being conducted.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Infant, children and adolescents who are aged 6 weeks to under 18 years or adult who are 18 years or older
2. Subjects who have been prescribed Prevenar 20 by their physician as per approved product label
3. Evidence of a personally signed and dated informed consent document indicating that the subject or their parent(s)/legal guardian, if applicable, have been informed of all pertinent aspects of the study

Exclusion Criteria:

Subjects meeting any of the following criteria will not be included in the study:

1. Subjects with contraindication according to approved label of Prevernar 20 (Pneumococcal 20-valent conjugate vaccine)
2. Any subjects (or a legally acceptable representative) who do not agree that Pfizer and companies working with Pfizer use his/her information

Min Age: 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population for this study is subjects aged 6 weeks or older who are determined to be administered Pneumococcal 20-valent conjugate vaccine according to the approved indications in routine clinical practice in Republic of Korea.
Sampling Method: Non-Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2025-11-28 (Estimated); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of solicited systemic reactions | From Day 1 through Day 7 after vaccination, where Day 1 is the day of vaccination
  The safety analysis set consists of all subjects who are prescribed Pneumococcal 20-valent conjugate vaccine by the investigator in the routine care, received at least one dose of Pneumococcal 20-valent conjugate vaccine according to the approved product label in Korea, and have at least one safety follow-up.
Frequency of solicited local reactions | From Day 1 through Day 10 after vaccination, where Day 1 is the day of vaccination
  The safety analysis set consists of all subjects who are prescribed Pneumococcal 20-valent conjugate vaccine by the investigator in the routine care, received at least one dose of Pneumococcal 20-valent conjugate vaccine according to the approved product label in Korea, and have at least one safety follow-up.
Frequency of Adverse Events (AEs) | 28 days after vaccination
  The safety analysis set consists of all subjects who are prescribed Pneumococcal 20-valent conjugate vaccine by the investigator in the routine care, received at least one dose of Pneumococcal 20-valent conjugate vaccine according to the approved product label in Korea, and have at least one safety follow-up.
Frequency of Adverse Events Special Interest (AESI) | 28 days after vaccination
  The safety analysis set consists of all subjects who are prescribed Pneumococcal 20-valent conjugate vaccine by the investigator in the routine care, received at least one dose of Pneumococcal 20-valent conjugate vaccine according to the approved product label in Korea, and have at least one safety follow-up.
Frequency of Adverse Drug Reactions (ADRs) | 28 days after vaccination
  The safety analysis set consists of all subjects who are prescribed Pneumococcal 20-valent conjugate vaccine by the investigator in the routine care, received at least one dose of Pneumococcal 20-valent conjugate vaccine according to the approved product label in Korea, and have at least one safety follow-up.
Frequency of Serious Adverse Events (SAEs) | 28 days after vaccination
  The safety analysis set consists of all subjects who are prescribed Pneumococcal 20-valent conjugate vaccine by the investigator in the routine care, received at least one dose of Pneumococcal 20-valent conjugate vaccine according to the approved product label in Korea, and have at least one safety follow-up.
Frequency of Serious Adverse Drug Reactions (SADRs) | 28 days after vaccination
  The safety analysis set consists of all subjects who are prescribed Pneumococcal 20-valent conjugate vaccine by the investigator in the routine care, received at least one dose of Pneumococcal 20-valent conjugate vaccine according to the approved product label in Korea, and have at least one safety follow-up.
Frequency of Unexpected AEs | 28 days after vaccination
  The safety analysis set consists of all subjects who are prescribed Pneumococcal 20-valent conjugate vaccine by the investigator in the routine care, received at least one dose of Pneumococcal 20-valent conjugate vaccine according to the approved product label in Korea, and have at least one safety follow-up.
Frequency of Unexpected ADRs | 28 days after vaccination
  The safety analysis set consists of all subjects who are prescribed Pneumococcal 20-valent conjugate vaccine by the investigator in the routine care, received at least one dose of Pneumococcal 20-valent conjugate vaccine according to the approved product label in Korea, and have at least one safety follow-up.
Frequency of Unexpected SAEs | 28 days after vaccination
  The safety analysis set consists of all subjects who are prescribed Pneumococcal 20-valent conjugate vaccine by the investigator in the routine care, received at least one dose of Pneumococcal 20-valent conjugate vaccine according to the approved product label in Korea, and have at least one safety follow-up.
Frequency of Unexpected SADRs | 28 days after vaccination
  The safety analysis set consists of all subjects who are prescribed Pneumococcal 20-valent conjugate vaccine by the investigator in the routine care, received at least one dose of Pneumococcal 20-valent conjugate vaccine according to the approved product label in Korea, and have at least one safety follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.